CLINICAL TRIAL: NCT01932528
Title: A Phase 1, Open-label, Non-randomised, Single-dose Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]-Telotristat Etiprate (LX1606) in Healthy Male Subjects
Brief Title: An Open-label Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]-Telotristat Etiprate in Males
Acronym: LX1606-104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-104-NRM
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoid Syndrome
Keywords: Absorption; Metabolism; Excretion
MeSH Terms: conditions — Serotonin Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 500 mg LX606 (Experimental): All subjects will receive a single oral 500 mg dose of [14C]-LX1606.
  Interventions: Drug: 500 mg [14C]-LX1606

INTERVENTIONS:
Drug: 500 mg [14C]-LX1606 — 500 mg dose of LX1606 containing a target dose of 3.32 Megabecquerel (MBq) of radiation as [14C]-LX1606.

SUMMARY:
To evaluate the metabolism and routes and extent of elimination of telotristat etiprate and its primary metabolite LX1033.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 30 to 65 years of age.
* Male subjects and their partners must agree to use an adequate method of contraception
* Historically able to produce a minimum of 1 bowel movement every day on most days

Exclusion Criteria:

* Female subjects
* Use of any medication or supplement within 5 days prior to Dosing
* Radiation exposure exceeding 5 millisieverts (mSv) in the last 12 months or 10 mSv in the last 5 years
* Current smokers or the use of cigarettes within 90 days prior to Screening
* History or renal disease or abnormal kidney function
* History of hepatic disease
* Acute diarrhea or constipation within 7 days of dosing
* Positive urine glucose at Screening

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of LX1606 and LX1033 | 7 days

SECONDARY OUTCOMES:
Time to maximum plasma concentration of and LX1033 | 7 days
Determination of total radioactivity in blood and plasma | 7 days
Mass balance recovery of total radioactivity in urine and feces | 7 days
Metabolite profiling and identification in plasma | 7 days
Metabolic profiling and identification in urine | 7 days
Metabolic profiling and identification in feces | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Doug Fleming, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Nottingham, United Kingdom